CLINICAL TRIAL: NCT01330693
Title: Cortical Excitability: Phenotype and Biomarker in ADHD Therapy
Brief Title: Cortical Excitability: Phenotype and Biomarker in Attention-deficit, Hyperactivity Disorder (ADHD) Therapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Cincinnati (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Floyd Sallee, Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R01MH081854-01A2 (NIH); 1R01MH081854-01A2 (NIH)
Record Dates: First submitted 2011-04-05; First posted 2011-04-07 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: ADHD; Atomoxetine; Biomarker
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atomoxetine (Active Comparator): Atomoxetine is FDA-approved for the treatment of ADHD symptoms in children
  Interventions: Drug: Atomoxetine
- Placebo (Placebo Comparator): Sugar pill
  Interventions: Drug: Sugar Pill

INTERVENTIONS:
Drug: Atomoxetine — Atomoxetine is FDA-approved for the treatment of ADHD symptoms in children. Single dose of 0.5 mg/kg at baseline visit. Then dose adjusted in an open-label design afterwards.
  Other Names: Strattera
  Arms: Atomoxetine
Drug: Sugar Pill — In-active sugar pill randomly assigned at baseline visit
  Arms: Placebo

SUMMARY:
The purpose of this study is to find out if children with attention-deficit, hyperactivity disorder (ADHD) have a difference in how their brain cells "fire" or react. The investigators also want to find if brain cell "firing" can tell us how severe of symptoms a child has from ADHD. Finally, the investigators want to see if giving an ADHD medication called atomoxetine can make the ADHD symptoms in a child better and if the improvement shows a change in brain "firing".

DETAILED DESCRIPTION:
This study will evaluate Short Interval Intracortical Inhibition (SICI) measured by pTMS as a marker of the hyperactive-impulsive dimension in 120 ADHD 7-12 years, medication-free children. This study will characterize the effects of a single dose of atomoxetine compared to placebo on cognitive correlates of SICI change. Participants will be randomized 2:1 to either atomoxetine or placebo. The study will also characterize the effects of four weeks of atomoxetine treatment on cortical inhibition and will correlate SICI change with clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent and assent
2. Meets DSM-IV criteria for ADHD, combined or inattentive subtype, based on K-SADS interview
3. Scores at least 1.5 SD higher than age and gender mean on ADHD RS, keyed to ADHD subtype (i.e., combined score for the combined subtype, inattentive subscale only for inattentive subtype, etc.)
4. Age: 7 - 12 years at study entry
5. Findings on physical exam, laboratory studies and ECG are judged to be normal for age and gender, as determined by study physician at study entry
6. There is not a co-existing medical condition for which TMS or ATX is contraindicated (for example pheochromocytoma).
7. Pulse and blood pressure within 95% of age and gender mean
8. Full scale IQ >75 (i.e., excluding mental retardation and the lower level of the borderline range)
9. Able to complete study instruments and swallow capsules
10. Willing to commit to the entire visit schedule for the study
11. No previous treatment with Atomoxetine
12. Must either be naive to ADHD study medication or not doing well on the current ADHD medication.

Exclusion Criteria:

1. Has one of the following exclusionary diagnoses: autism/ pervasive developmental disorder, mental retardation, schizophrenia, a psychotic disorder, bipolar disorder, severe depressive or conduct disorder
2. Has a comorbid disorder that is otherwise allowable, but which requires a treatment that is not being offered in the study, and should be the primary focus of treatment, in the opinion of the PI
3. Has a medical or neurologic disorder that would preclude taking the ATX, or which would potentially confound the assessment of ADHD and/or TMS outcomes, in the opinion of the PI (for example pheochromocytoma, or for specific purposes of this study uncontrolled seizure disorder or organic brain syndrome).
4. Taking a systemic medication which might interfere with the metabolism or efficacy assessment of ATX in this study
5. History of allergic reactions to multiple medications
6. History of alcohol or drug abuse in the past 3 months Has been in a medication treatment study in the past 30 days
7. Females of childbearing age who are sexually active, do not use acceptable birth control (double barrier method), or are not abstinent. Abstinence is defined as no sexual activity for at least 3 months before the start of the study and the intention to abstain from sexual activity during the study period). Double barrier methods allowed include: condoms or diaphragms combined with spermicide use, intrauterine devices (IUD), and oral, transdermal, injectable or implantable hormonal medications (Ortho-Evra, Norplant, Depo-Provera, and similar prescription products) for at least one month before entering the study and continuing its use throughout the study. Birth control pills alone are not acceptable forms of birth control for this study.
8. Has any prior neurological condition that might increase the risk of an adverse event with TMS. For the purpose of this study we are excluding children with a current or prior history of epilepsy.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2009-09; Primary Completion 2015-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Efficacy outcome as change from baseline in ADHDRS total score | At 4 weeks
SICI as a marker of ADHD Behaviors | Baseline visit
  To evaluate pTMS-evoked Short Interval Cortical Inhibition (SICI) as a marker of the hyperactive-impulsive dimension in Attention Deficit Hyperactivity Disorder
Cognitive Correlates of SICI Change | 2 hours (at baseline visit)
  To determine cognitive correlates of SICI change, the study will first measure SICI at at rest and concurrently during the Stop-task. This process will then be repeated 2 hours after a single dose (0.5 mg/kg) of atomoxetine (ATX) or placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Floyd R Sallee, MD, Principal Investigator — University of Cincinnati
Locations (2):
- United States (2):
  - University of Cincinnati, Cincinnati, Ohio
  - Cincinnati Children's Hospital, Cincinnati, Ohio